CLINICAL TRIAL: NCT01536379
Title: BEL114424: A Phase 2 Pilot, Multicentered, Randomised, Double Blind, Placebo-Controlled Study to Evaluate the Potential for Efficacy and the Safety of Belimumab Plus Standard of Care Versus Placebo Plus Standard of Care in the Prevention of Allograft Rejection in Adult Subjects After Renal Transplantation
Brief Title: A Study of Belimumab in the Prevention of Kidney Transplant Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114424
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Transplantation, Organ
Keywords: Infection; Quality of Life
MeSH Terms: conditions — Infections | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belimumab 10 mg (Experimental): Subjects will receive belimumab 10 mg/ Kilogram (kg) infusion on Days 0, 14, 28 and every 4 weeks thereafter for a total of 7 infusions. The last dose of investigational product will be administered at the Week 20 visit; In addition to investigational product, all subjects will receive standard of care.
  Interventions: Drug: Belimumab
- Placebo (Placebo Comparator): Subjects will receive placebo infusion on Days 0, 14, 28 and every 4 weeks thereafter for a total of 7 infusions. The last dose of investigational product will be administered at the Week 20 visit; In addition to investigational product, all subjects will receive standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belimumab — Belimumab (10 mg/kg) will be given as an intravenous solution over a 1 hour time period administered every 4 weeks for 24 weeks (with an additional dose at Week 2)
  Arms: Belimumab 10 mg
Drug: Placebo — Placebo will be given as an intravenous solution over a 1 hour time period administered every 4 weeks for 24 weeks (with an additional dose at Week 2)
  Arms: Placebo

SUMMARY:
Kidney transplantation is the best treatment for many patients with kidney failure. Sometimes a transplanted kidney is rejected by the patient's immune system. Many types of immune system cells, including B cells, are active in rejection. B cells produce antibodies against anything the body sees as non-self, like germs or a transplanted kidney. Most medicines that help prevent transplant rejection affect cells other than B cells. Belimumab is a medication used to treat a disease called lupus. Belimumab slows development of antibody-producing B cells. This study will test whether belimumab works on parts of the immune system that cause rejection. Twenty to thirty adults getting a kidney transplant will be in this study. Like flipping a coin, a computer will randomly assign half to be given belimumab and half to be given placebo (a fake medicine). Patients and doctors will not know which medicine was assigned until the study is over. A total of 7 doses of study medicine will be given through a vein. One dose will be given during transplant surgery, and the other 6 will be given 2, 4, 8, 12, 16 and 20 weeks after transplant surgery. Usual transplant medicines will also be given. After all of the doses have been given, patients will be watched and tested at 24, 36, and 52 weeks after the transplant surgery. Blood samples will be tested to see what study medicines do to the immune system in transplant patients. If patients get a kidney biopsy, the samples will be tested to see if belimumab had any effect. Patients will be asked many questions to see if they are having any side effects. The study will be done at Addenbrooke's Hospital in Cambridge and Guys &St Thomas Hospital in London, United Kingdom. A pharmaceutical company, GlaxoSmithKline, is funding the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for kidney transplantation: Considered eligible for transplantation after undergoing multidisciplinary evaluation at the institution at which the transplantation will be performed
* Donor characteristics: Receiving a deceased donor kidney or a living donor kidney allograft
* Age & Gender: Male or female between 18 and 75 years of age, inclusive, at the time of signing the informed consent
* Female Subjects: Not pregnant or nursing and at least one of the following conditions apply: a. Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea. In the absence of confirmatory laboratory assessments [(a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 million international units per milliliter (MIU/mL) and estradiol < 40 picogram per milliliter (pg/mL) (<147 picomole per liter [pmol/L])] in questionable cases, female subjects will be required to use one of the contraception methods as described by the investigator or designee, until confirmatory results become available; b. Questionable post-menopausal status and agrees to use one of the contraception methods as described by the investigator or designee, from Day 0 until 16 weeks after the last dose of investigational product or until postmenopausal status is confirmed with a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MIU/mL and estradiol status who are using hormone replacement therapy (HRT) will be required to use one of the contraception methods as described by the investigator or designee, until post-menopausal status is confirmed. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; c. Child-bearing potential and agrees to use one of the contraception methods as described by the investigator or designee, from Day 0 until 16 weeks after the last dose of investigational product.
* Liver function (most recent values available before transplantation): alanine aminotransferase (ALT) < 2x upper limit of normal (ULN); bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Immunosuppressants: at the time of transplantation, planned to receive a combination of immunosuppressants including basiliximab, mycophenolate mofetil, tacrolimus, prednisolone

Exclusion Criteria:

* Donor characteristics: receiving a kidney allograft from a donor with any of the following characteristics: a) cold ischemic time exceeding 36 hours; b) age < 5 years old; c) for donors after brain death (DBD), age >70 years old; d) for donors after cardiac death (DCD) age >70 years old; e) ABO blood type incompatible against the recipient; f) 0 0 0 HLA-A -B -DR mismatch against the recipient by National Health Service Blood and Transplant (NHSBT criteria; g) T- and/or B-cell positive crossmatch by complement dependent cytotoxicity or flow cytometry against the recipient. Note :- (In some situations it may be that a pre-existing T- and/or B-cell positive crossmatch by complement dependent cytotoxicity or flow cytometry against the recipient will only be fully revealed immediately after the transplant; in such situations they will be recorded as having met exclusion criteria and withdraw from further involvement in the study; h) serology positive for hepatitis B (except hepatitis B surface antibody and prior vaccination), hepatitis C or human immunodeficiency virus (HIV)
* Transplant other than kidney: has previously received a hematopoietic stem cell/marrow transplant or an organ transplant other than a kidney (with the exception of corneal transplantation)
* Planned immunosuppressant regimen: are being considered for steroid-free or alemtuzumab induction
* Prior therapy at any time: has ever received any of the following: a) B-cell targeted therapy (e.g., rituximab, other anti-CD20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], TACI fragment, crystallizable (Fc), or belimumab)
* 364 Day prior therapy: has received any of the following within 364 days before Day 0: a) Cyclophosphamide; b) Abatacept; c) A biologic investigational agent other than B-cell targeted therapy [e.g., abetimus sodium, anti CD40L antibody (e.g., BG9588/ IDEC 131; investigational agent applies to any drug not approved for sale in the country in which it is being used]
* 90 Day prior therapy: has received any of the following within 90 days before Day 0: a) Anti- Tumor necrosis factor (TNF) or anti-Interleukin (IL)-6 therapy (e.g., adalimumab, etanercept, infliximab, tocilizumab); b) Interleukin-1 receptor antagonists (e.g., anakinra); c) Intravenous immunoglobulin (IVIG); d) Plasmapheresis, leukapheresis
* 60 Day prior therapy: has received any of the following within 60 days before Day 0: a) A non-biologic investigational agent (investigational agent applies to any drug not approved for sale in the country in which it is being used); b) Any new immunosuppressive/immunomodulatory agent; tacrolimus, Mycophenolate mofetil (MMF), and corticosteroids are permitted. Inhaled steroids and new topical immunosuppressive agents (e.g., eye drops, topical creams) are also allowed.
* 30 Day prior therapy: has received any of the following within 30 days before Day 0: a) A live vaccine; b) An increase in dose of an immunosuppressive/immunomodulatory agent (decreases in dose or discontinuations are permitted). Increases in doses of tacrolimus, MMF, and corticosteroids are permitted.
* Malignancy: has a history of malignancy in the past 5 years except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Acute or chronic infection: has required management of acute or chronic infections (excludes prophylaxis of infections), as follows: a) Currently receiving any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria), which, in the opinion of the investigator, could put the subject at undue risk; b) Hospitalized for treatment of infection within 30 days before Day 0, which, in the opinion of the investigator, could put the subject at undue risk ; c) Treated for an infection with parenteral (intravenous or intramuscular)] antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 30 days before Day 0, which, in the opinion of the investigator, could put the subject at undue risk
* Other disease/conditions: has any of the following: a) clinical evidence of significant unstable or uncontrolled acute or chronic diseases (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk; b) a surgical procedure planned in the 6 months after Day 0, other than kidney transplantation or related procedure; c) a known history of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the investigator, makes the subject unsuitable for the study
* Hepatitis: known to have serologic evidence of hepatitis B infection based on the results of testing for hepatitis B surface antigen (HBsAg), or antibodies against hepatitis B core antigen (HBc) and/or hepatitis B surface antigen (HBs) as follows: a) Patients positive for HBsAg are excluded; ) Patients negative for HBsAg and anti-HBc antibody but positive for anti-HBs antibody and with no history of hepatitis B vaccination are excluded; c) Patients negative for HBsAg but positive for both anti-HBc and anti-HBs antibodies are excluded; d) Patients negative for HBsAg and anti-HBs antibody but positive for anti-HBc antibody are excluded; e) Or has known serologic evidence of hepatitis C infection based on the results of testing for hepatitis C antibody and hepatitis C recombinant immunoblot assay (RIBA) as follows: Patients with a positive test for Hepatitis C antibody confirmed on the same sample with a Hepatitis C RIBA immunoblot assay. Patients who are positive for Hepatitis C antibody, and who are negative when the Hepatitis C RIBA immunoblot assay is performed on the same sample, will be eligible to participate. Patients who are positive for Hepatitis C antibody and who have a positive or indeterminate result when the Hepatitis C RIBA immunoblot assay is performed on the same sample, will not be eligible to participate.
* HIV: known to have a historically positive HIV test or tests positive at screening for HIV.
* Immunodeficiency: recipient with a history of immunodeficiency (defined as Immunoglobulin A isotype (IgA) level <10 milligrams per deciliter (mg/dL) or have Immunoglobulin G isotype (IgG) level <400 mg/dL).
* Laboratory abnormalities: has an abnormal laboratory assessment, which is judged clinically significant by the investigator.
* Lymphopenia: has a lymphocyte count <500/ millimeter (mm)^3.
* Drug Sensitivity: has a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy including a previous anaphylactic reaction to parenteral administration contrast agents, human or murine proteins or monoclonal antibodies that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Substance abuse: has evidence of current drug or alcohol abuse or dependence.
* Blood donation: where participation in the study would result in donation of blood or blood products in excess of 700 mL within a 56-day period
* Venous access: has venous access limitations likely to preclude monthly infusions
* Compliance: is unlikely to comply with scheduled study visits based on investigator judgment or has a history of substance abuse, psychiatric disorder or condition that may compromise communication with the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Banham GD, Flint SM, Torpey N, Lyons PA, Shanahan DN, Gibson A, Watson CJE, O'Sullivan AM, Chadwick JA, Foster KE, Jones RB, Devey LR, Richards A, Erwig LP, Savage CO, Smith KGC, Henderson RB, Clatworthy MR. Belimumab in kidney transplantation: an experimental medicine, randomised, placebo-controlled phase 2 trial. Lancet. 2018 Jun 30;391(10140):2619-2630. doi: 10.1016/S0140-6736(18)30984-X. Epub 2018 Jun 14. PMID 29910042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 renal transplant recipients were enrolled, of which 28 were randomized and 25 were transplanted.
Pre-assignment Details: Participants were randomized to 1 of the 2 treatments groups in a 1:1 ratio and received standard of care in addition to investigational products (IPs). Participants received IP infusion on Day 0, Day 14, Day 28 and every 4 weeks thereafter for a total of 7 infusions.
Groups:
- Placebo: Participants received normal saline (0.9% sodium chloride) via intravenous infusion over 1 hour, every 4 weeks for 24 weeks (with an additional dose at week 2) in addition to standard of care assessments, treatment and other interventions according to institutional protocols from the time of transplantation throughout the study.
- Belimumab 10mg/kg: Participants received 10 milligram (mg) /kilogram (kg) belimumab in 250 milliliter (mL) normal saline via intravenous infusion over 1 hour, every 4 weeks for 24 weeks (with an additional dose at week 2) standard of care assessments, treatment and other interventions according to institutional protocols from the time of transplantation throughout the study.
Period: Overall Study
Arm/Group | Placebo | Belimumab 10mg/kg
Started | 13 | 12
Completed | 11 | 9
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab 10mg/kg | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.0 (14.02) | 54.3 (11.02) | 52.6 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 9 | 5 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 12 | 11 | 23
  Asian | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in naïve B Cells From Baseline to Week 24
Description: Naive B cell is cell that is not exposed to antigen. Naïve B cell count is CD20+CD27 concentration of cells (conc-cell)/cubic millimeter (cumm). Change from Baseline in naïve B cells was calculated as the value at Week 24 minus the value at Baseline. MITT Population consisted of all participants randomized to treatment, who have had taken at least one dose of study. Participants analyzed included those who had data at Week 24 for naïve B cells count (MITT Population). Baseline value used in the analysis was of Day 0 (Day of transplant). Adjusted mean differences (treatment-placebo) and 95% confidence intervals for differences were obtained from mixed-models repeated-measures (MMRM) model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments.
Time Frame: Baseline and Week 24
Population: Modified Intent to treat (MITT) Population
Measure: Least Squares Mean (Standard Error); unit: cells/mm^3
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 9 | 7
cells/mm^3 | 4.0 (25.55) | -30.4 (27.50)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -34.4, 95% CI 2-sided [-109.5 to 40.7], Standard Error of Mean 37.24

2. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)
Description: Number of participants with AEs, SAEs and AESI are summarized. The On-treatment (OT) phase started on the day and time of receiving the start of the first infusion and ended on the last dose date plus 28 days. The Post-treatment (PT) phase started 29 days after day of last dose up to 1 year. An AE is any untoward medical occurrence, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that at any dose results in, death, is life threatening, Requires hospitalization or prolongation of existing hospitalization, Results in disability/incapacity, Is a congenital anomaly/birth defect or event that but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed. AESI included malignant neoplasms, infusion/anaphylaxis/hypersensitivity reactions, all infections, depression/suicide/self-injury, deaths.
Time Frame: Up to 1 year
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Participants
  OT AEs | 10 | 11
  PT AEs | 9 | 10
  OT SAEs | 7 | 5
  PT SAEs | 2 | 2
  Malignant neoplasms | 0 | 0
  Post-Infusion Systemic Reactions | 0 | 1
  All Infections | 6 | 7
  Depression/suicide/self-injury | 0 | 0
  Deaths | 1 | 0

3. Primary Outcome: Number of Incidence of All Infections and Serious Infections
Description: All infections included: 1. Opportunistic infections per-clinical assessment, 2. Herpes Zoster, a. Recurrent, b. Disseminated, 3. Sepsis. Opportunistic infections were identified using list of preferred terms as per Medical Dictionary for Regulatory Activities (MedDRA) version 18.1. Any events falling under these preferred terms were adjudicated to determine if criteria was met for an opportunistic infection.
Time Frame: Up to 1 year
Population: mITT Population
Measure: Number; unit: Infections
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Infections
  All Infections | 8 | 7
  Serious Infections | 2 | 1
  All Opportunistic Infections | 7 | 5
  Serious Opportunistic Infections | 1 | 0
  All Herpes Zoster | 0 | 1
  Serious Herpes Zoster | 0 | 0
  Sepsis | 3 | 2
  Serious Sepsis | 2 | 1

4. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 24 and Week 52
Description: Change from Baseline in SBP and DBP were assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value at Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
millimeter of mercury (mmHg)
  DBP Week 24; n=9, 7 | -4.444 (14.3275) | 7.286 (13.8289)
  DBP Week 52; n=11, 10 | -6.545 (13.9668) | 4.200 (8.5479)
  SBP Week 24; n=9, 7 | 2.000 (26.0960) | 10.000 (35.9444)
  SBP Week 52; n=11, 10 | -2.909 (27.2046) | 3.300 (27.9008)

5. Primary Outcome: Change From Baseline in Heart Rate From Baseline at Week 24 and Week 52
Description: Change from Baseline in heart rate was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value at Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Beats per minute (BPM)
  Week 24; n=8, 6 | 5.125 (16.8983) | 1.500 (13.6345)
  Week 52; n=11, 9 | 2.000 (11.5065) | -2.444 (15.4200)

6. Primary Outcome: Change From Baseline in Body Temperature From Baseline at Week 24 and Week 52
Description: Change from Baseline in body temperature was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value at Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Degree Centigrade
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Degree Centigrade
  Week 24; n=8, 6 | 0.025 (0.7025) | -0.233 (0.5007)
  Week 52; n=11, 10 | -0.045 (0.4803) | 0.030 (0.5417)

7. Primary Outcome: Number of Participants Outside the Normal Range (NR) for SBP and DBP at Week 24 and Week 52
Description: Number of participants outside the normal range (NR) for SBP and DBP was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Number of participants outside the normal range are summarized by less than (<) normal range and greater than (>) normal range categories at Week 24 and Week 52. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Participants
  DBP, > NR, Week 24; n=9, 7 | 1 | 1
  DBP, < NR, Week 24; n=9, 7 | 1 | 2
  DBP, > NR, Week 52; n=11, 10 | 3 | 0
  DBP, < NR, Week 52; n=11, 10 | 2 | 1
  SBP, > NR, Week 24; n=9, 7 | 5 | 3
  SBP, < NR, Week 24; n=9, 7 | 0 | 0
  SBP, > NR, Week 52; n=11, 10 | 5 | 4
  SBP, < NR, Week 52; n=11, 10 | 0 | 1

8. Primary Outcome: Number of Participants Outside the Normal Range (NR) for Heart Rate at Week 24 and Week 52
Description: Number of participants outside the normal range (NR) for heart rate was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Number of participants outside the normal range are summarized by less than (<) normal range and greater than (>) normal range categories at Week 24 and Week 52. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Participants
  > NR Week 24; n=8, 6 | 1 | 0
  < NR Week 24; n=8, 6 | 2 | 0
  > NR Week 52; n=11, 9 | 0 | 0
  < NR Week 52; n=11, 9 | 1 | 1

9. Primary Outcome: Number of Participants Outside the Normal Range (NR) for Body Temperature at Week 24 and Week 52
Description: Number of participants outside the normal range (NR) for body temperature was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Number of participants outside the normal range are summarized by less than (<) normal range and greater than (>) normal range categories at Week 24 and Week 52. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Participants
  > NR Week 24; n=8, 6 | 0 | 0
  < NR Week 24; n=8, 6 | 3 | 4
  > NR Week 52; n=11, 10 | 0 | 0
  < NR Week 52; n=11, 10 | 5 | 2

10. Primary Outcome: Change From Baseline in the Indicated Hematology Parameters at Week 24 and Week 52
Description: Hematology parameters included: basophils (B), eosinophils (E), lymphocytes (L), monocytes (M), total neutrophils (N), platelet count (PC) and white blood cells (WBC). Change from Baseline in haematology parameter was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Gills/Liter (GI/L)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Gills/Liter (GI/L)
  B Week 24; n=9, 6 | -0.001 (0.0215) | -0.015 (0.0207)
  B Week 52; n=10, 10 | 0.033 (0.1024) | -0.005 (0.0357)
  E Week 24; n=9, 6 | -0.531 (1.0250) | -0.140 (0.1274)
  E Week 52; n=10, 10 | -0.392 (0.8048) | -0.127 (0.1489)
  L Week 24; n=9, 6 | -0.218 (0.6457) | -0.347 (0.3467)
  L Week 52; n=10, 10 | 0.085 (0.5841) | -0.245 (0.3357)
  M Week 24; n=9, 6 | -0.097 (0.2231) | -0.365 (0.3509)
  M Week 52; n=10, 10 | 0.001 (0.1799) | -0.111 (0.3892)
  TN Week 24; n=9, 6 | 0.946 (2.6602) | -0.083 (2.4752)
  TN Week 52; n=10, 10 | 1.657 (3.5533) | -0.606 (3.3406)
  PC Week 24; n=9, 6 | 15.9 (59.64) | 7.3 (40.35)
  PC Week 52; n=11, 10 | 18.1 (55.81) | -10.0 (54.14)
  WBC Week 24; n=9, 6 | 0.10 (3.483) | -0.95 (2.868)
  WBC Week 52; n=11, 10 | 1.47 (3.572) | -1.11 (3.557)

11. Primary Outcome: Change From Baseline in the Haematology Parameter- Hemoglobin at Week 24 and Week 52
Description: Change from Baseline in hemoglobin was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Grams per Liter (G/L)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Grams per Liter (G/L)
  Week 24; n=9, 6 | 5.4 (24.84) | 13.2 (28.90)
  Week 52; n=11, 10 | 12.6 (22.69) | 6.3 (23.48)

12. Primary Outcome: Change From Baseline in the Hematology Parameter- Hematocrit at Week 24 and Week 52
Description: Endpoint was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Percentage of blood
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Percentage of blood
  Week 24; n=9, 6 | 0.0216 (0.06625) | 0.0477 (0.09540)
  Week 52; n=11, 10 | 0.0434 (0.06813) | 0.0238 (0.07045)

13. Primary Outcome: Change From Baseline in Haematology Parameter- Mean Corposcular Hemoglobin (MCH) at Week 24 and Week 52
Description: Change from Baseline in MCH was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Picogram (pg)
  Week 24; n=8, 6 | -0.79 (2.173) | -1.37 (2.683)
  Week 52; n=10, 10 | -1.59 (1.516) | -1.93 (2.743)

14. Primary Outcome: Change From Baseline in Haematology Parameter- Mean Corposcular Volume (MCV) at Week 24 and Week 52
Description: Change from Baseline in MCV was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Femtoliter (FL)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Femtoliter (FL)
  Week 24; n=9, 6 | -1.73 (6.430) | -2.55 (8.198)
  Week 52; n=11, 10 | -3.58 (4.340) | -4.61 (7.041)

15. Primary Outcome: Change From Baseline in Haematology Parameter- Red Blood Cell (RBC) at Week 24 and Week 52
Description: Change from Baseline in RBC was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Tera (TI)/L
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Tera (TI)/L
  Week 24; n=9, 6 | 0.298 (0.6716) | 0.645 (0.8097)
  Week 52; n=11, 10 | 0.635 (0.7064) | 0.468 (0.5884)

16. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter- Albumin at Week 24 and Week 52
Description: Change from Baseline in albumin was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
G/L
  Week 24; n=9, 7 | 4.1 (2.62) | 2.9 (4.91)
  Week 52; n=10, 10 | 2.9 (3.00) | 1.8 (4.98)

17. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter- ALP, ALT, AST at Week 24 and Week 52
Description: Clinical chemistry parameter included alkaline phosphatase (ALP), alanine amino Transferase (ALT) and aspartate amino transferase (AST). Endpoint was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: International Unit (IU)/L
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
International Unit (IU)/L
  ALP Week 24; n=9, 7 | -16.0 (26.14) | -5.0 (60.03)
  ALP Week 52; n=10, 10 | -17.5 (35.25) | 19.9 (80.63)
  ALT Week 24; n=9, 7 | 1.0 (15.86) | 5.1 (7.56)
  ALT Week 52; n=10, 10 | -2.5 (11.16) | 2.1 (5.80)
  AST Week 24; n=6, 3 | 3.2 (7.91) | 7.3 (4.04)
  AST Week 52; n=7, 4 | 3.3 (5.68) | 9.3 (3.86)

18. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter- Direct Bilirubin, Total Bilirubin and Creatinine at Week 24 and Week 52
Description: Clinical chemistry parameters included direct bilirubin (DB), total bilirubin (TB) and creatinine (C). Endpoint was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Micromole per Liter (umol/L)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Micromole per Liter (umol/L)
  DB Week 24; n=8, 3 | 0.6 (1.51) | -0.7 (3.06)
  DB Week 52; n=9, 5 | 0.9 (1.54) | 0.2 (1.30)
  TB Week 24; n=9, 7 | 3.0 (6.50) | 2.7 (5.22)
  TB Week 52; n=10, 10 | 2.9 (5.26) | 2.9 (3.38)
  C Week 24; n=9, 7 | -471.1 (317.54) | -571.3 (183.53)
  C Week 52; n=10, 10 | -468.4 (310.54) | -609.8 (271.89)

19. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter- Ca, CO2/Bicar, Gl, K, Na, PhI, U/BUN at Week 24 and Week 52
Description: Clinical chemistry parameters included calcium (Ca), carbon dioxide content/bicarbonate (CO2/Bicar), glucose (Gl), potassium (K), sodium (Na), phosphorus inorganic (PhI), urea/blood urine nitrogen (U/BUN). Endpoint was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Millimole (MMOL)/L
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Millimole (MMOL)/L
  Ca Week 24; n=9, 7 | 0.116 (0.1344) | 0.167 (0.1942)
  Ca Week 52; n=10, 9 | 0.116 (0.1013) | 0.128 (0.1386)
  CO2/Bicar Week 24; n=7, 6 | -3.73 (5.951) | 1.70 (3.449)
  CO2/Bicar Week 52; n=8, 9 | -2.68 (5.142) | 0.77 (3.588)
  Gl Week 24; n=5, 5 | 0.20 (3.093) | -0.04 (2.003)
  Gl Week 52; n=5, 8 | -0.32 (2.483) | 1.79 (4.107)
  K Week 24; n=9, 7 | 0.06 (0.723) | -0.63 (0.923)
  K Week 52; n=10, 10 | -0.02 (0.535) | -0.44 (0.877)
  Na Week 24; n=9, 7 | -0.6 (4.03) | 5.9 (5.01)
  Na Week 52; n=10, 10 | -0.7 (3.71) | 2.2 (4.71)
  PhI Week 24; n=8, 7 | -0.225 (0.3843) | -0.913 (0.5862)
  PhI Week 52; n=9, 9 | -0.227 (0.4234) | -0.726 (0.5453)
  U/BUN Week 24; n=9, 6 | -5.91 (12.164) | -9.47 (9.128)
  U/BUN Week 52; n=10, 9 | -8.13 (14.967) | -9.01 (7.323)

20. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter- Glomerular Filtration Rate (GFR) at Week 24 and Week 52
Description: Change from Baseline in GFR was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: milliliter (mL)/Minute (min)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
milliliter (mL)/Minute (min)
  Week 24; n=9, 7 | 42.80 (23.604) | 44.36 (10.731)
  Week 52; n=10, 10 | 42.33 (29.140) | 53.75 (15.176)

21. Primary Outcome: Change From Baseline in Immunoglobulin A (IgA), Immunoglobulin G (IgG) and Immunoglobulin M (IgM) at Week 24 and Week 52
Description: Change from Baseline in immunoglobulins IgA, IgG and IgM was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Change from Baseline was calculated as the value on Week 24 and Week 52 minus the value at Baseline. Baseline value used in the analysis was of Day 0 (Day of transplant). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
G/L
  IgA Week 24; n=2, 3 | -0.500 (0.2828) | -0.433 (0.6429)
  IgA Week 52; n=2, 3 | -0.300 (0.0000) | -0.500 (0.5292)
  IgG Week 24; n=6, 6 | -1.02 (1.184) | -2.40 (1.731)
  IgG Week 52; n=10, 9 | 0.78 (3.595) | -2.13 (1.702)
  IgM Week 24; n=2, 3 | -0.100 (0.0000) | -0.133 (0.3512)
  IgM Week 52; n=2, 3 | 0.0000 (0.0000) | -0.333 (0.4933)

22. Secondary Outcome: Median Percent Change From Baseline in Memory B Cell Count at Week 24 and Week 52
Description: Memory B cells are B cell sub-type that are formed within germinal centres following primary infection and are important in generating an accelerated and more robust antibody-mediated immune response in the case of re-infection. Memory B cell count included CD20+CD27+ cells/mm^3. Baseline value used in the analysis was of Day 0 (Day of transplant). Endpoint was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Percent change from Baseline in Memory B cell count was calculated as the value at Week 24 and Week 52 minus the value at Baseline multiplied by 100. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Median Difference and 95% confidence interval of difference obtained using the Hodges-Lehmann method.
Time Frame: Baseline, Week 24 and Week 52
Population: mITT Population
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Percent change
  Week 24; n=9, 7 | -12.5 [-88 to 320] | 177.8 [40 to 800]
  Week 52; n=10, 7 | 2.4 [-67 to 340] | -33.3 [-80 to 44]
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Median Difference (Final Values) = 204.35, 95% CI 2-sided [90.00 to 550.00] — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Median Difference (Final Values) = -33.06, 95% CI 2-sided [-169.84 to 25.00] — Week 52 comparison

23. Secondary Outcome: Activated Memory B Cells Count at Week 24 and Week 52
Description: Activated memory B cell-CD95% count is CD19+CD27+CD95 conc-cells/mL. Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: cells/mL
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
cells/mL
  Week 24; n=9, 7 | 37157.2 (16664.42) | 38389.6 (18682.83)
  Week 52; n=10, 8 | 24220.8 (15744.17) | 11092.5 (17711.36)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = 1232.40, 95% CI 2-sided [-50457.0 to 52921.8], Standard Error of Mean 25735.56 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -13128.35, 95% CI 2-sided [-61868.9 to 35612.2], Standard Error of Mean 24165.18 — Week 52 comparison

24. Secondary Outcome: Activated Memory B Cells Percentage at Week 24 and Week 52
Description: Activated memory B cell-CD95% percentage is CD19+CD27+CD95+ (%CD19/CD27). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of activated memory B cells
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Percentage of activated memory B cells
  Week 24; n=9, 7 | 32.8 (5.94) | 19.0 (6.06)
  Week 52; n=11, 10 | 32.0 (5.07) | 38.8 (5.48)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -13.8, 95% CI 2-sided [-31.3 to 3.7], Standard Error of Mean 8.78 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-8.6 to 22.2], Standard Error of Mean 7.68 — Week 52 comparison

25. Secondary Outcome: Transitional B Cells Count at Week 24 and Week 52
Description: Transitional B cell count (Newell) is CD19+CD24b+CD38b+IgD+ (Conc-cells/mL). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: cells/mL
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
cells/mL
  Week 24; n=9, 7 | 5470 (2910.9) | 2679 (3518.4)
  Week 52; n=10, 8 | 7110 (2836.7) | 6652 (3291.5)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -2791, 95% CI 2-sided [-12105 to 6524], Standard Error of Mean 4651.1 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -458, 95% CI 2-sided [-9487 to 8572], Standard Error of Mean 4501.8 — Week 52 comparison

26. Secondary Outcome: Transitional B Cells Percentage at Week 24 and Week 52
Description: Transitional B cell percentage (Newell) is CD19+CD24b+CD38b+IgD+ (%CD19+). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of transitional B cells
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Percentage of transitional B cells
  Week 24; n=9, 7 | 2.43 (0.776) | 1.14 (0.869)
  Week 52; n=11, 10 | 2.61 (0.713) | 3.41 (0.731)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-3.59 to 1.01], Standard Error of Mean 1.156 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-1.24 to 2.82], Standard Error of Mean 1.017 — Week 52 comparison

27. Secondary Outcome: Activated T Cell Count at Week 24 and Week 52
Description: A T cell is a type of lymphocyte that plays a central role in cell-mediated immunity. Activated T cell count Codarri is CD4+ CD25hi CD45RA- IL 7Rhi (Conc-cells/mL). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: cells/mL
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
cells/mL
  Week 24; n=9, 6 | 109279.5 (22998.02) | 78952.7 (26155.19)
  Week 52; n=10, 7 | 122304.7 (21898.24) | 75349.4 (24313.62)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -30326.9, 95% CI 2-sided [-100559.1 to 39905.3], Standard Error of Mean 34677.86 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -46955.3, 95% CI 2-sided [-113218.9 to 19308.3], Standard Error of Mean 32594.81 — Week 52 comparison

28. Secondary Outcome: Activated T Cell Percentage at Week 24 and Week 52
Description: Activated T cell percentage (Codarri)= CD4+ CD25hi CD45RA- IL 7Rhi (% of CD4+). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of activated T cell
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Percentage of activated T cell
  Week 24; n=9, 6 | 17.0 (2.29) | 14.0 (2.58)
  Week 52; n=10, 7 | 15.2 (2.15) | 14.7 (2.33)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-10.1 to 4.2], Standard Error of Mean 3.54 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-7.2 to 6.3], Standard Error of Mean 3.35 — Week 52 comparison

29. Secondary Outcome: Regulatory T Cell Count at Week 24 and Week 52
Description: Regulatory T cell count is CD4+ CD25hi IL-7Rlo (Conc-cells/mL). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: cells/mL
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
cells/mL
  Week 24; n= 9, 7 | 23586.2 (8427.77) | 24234.5 (9238.41)
  Week 52; n= 10, 8 | 33038.7 (7676.99) | 27419.8 (9093.84)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = 648.3, 95% CI 2-sided [-24661.1 to 25957.7], Standard Error of Mean 12618.44 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -5618.9, 95% CI 2-sided [-29994.8 to 18757.0], Standard Error of Mean 12153.03 — Week 52 comparison

30. Secondary Outcome: Regulatory T Cell (%CD4) at Week 24 and Week 52
Description: Regulatory T cell (%CD4) = CD4+ CD25hi IL-7Rlo (% of CD4+). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of Regulatory T cell
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Percentage of Regulatory T cell
  Week 24; n= 9, 7 | 4.4 (1.12) | 4.6 (1.25)
  Week 52; n= 11, 10 | 5.0 (1.01) | 4.4 (1.04)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-3.2 to 3.5], Standard Error of Mean 1.67 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-3.5 to 2.3], Standard Error of Mean 1.45 — Week 52 comparison

31. Secondary Outcome: Mean Activated: Regulatory T Cell Ratio at Week 24 and Week 52
Description: Activated: regulatory T cell ratio is Activated T cell CD4+CD25hi CD45RA IL 7Rhi (absolute number)/ Regulatory T cell CD4+CD25hi CD45RA IL 7Rlo (absolute number). Adjusted mean difference (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Ratio
  Week 24; n= 9, 6 | 4.88 (0.832) | 3.33 (0.915)
  Week 52; n= 10, 7 | 4.62 (0.779) | 3.61 (0.942)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-4.07 to 0.98], Standard Error of Mean 1.255 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-3.68 to 1.67], Standard Error of Mean 1.329 — Week 52 comparison

32. Secondary Outcome: Proportion of Participants With Episodes of Acute Rejection at Week 24 and Week 52
Description: The endpoint diagnosis was made by a proven biopsy result. Number of rejections only counted once per participant. The proportion of participants with episodes of acute rejection was assessed at Week 24 (at the end of therapy) and at Week 52 (at study end). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population. Participants analyzed had at least one biopsy.
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
Proportion of participants
  Week 24; n=5, 6 | 0.4 | 0.33
  Week 52; n=5, 6 | 0.6 | 0.33
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Difference in Proportion = -0.067, 95% CI 2-sided [-0.638 to 0.505] — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Difference in Proportion = -0.267, 95% CI 2-sided [-0.838 to 0.305] — Week 52 comparison

33. Secondary Outcome: Mean Serum Creatinine at Week 24 and Week 52
Description: Adjusted mean difference for serum creatinine values (treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction, at Week 24 and Week 52. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: micromole/L
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
micromole/L
  Week 24; n=9, 7 | 115.1 (35.24) | 112.3 (38.20)
  Week 52; n= 10, 10 | 135.4 (33.50) | 122.6 (33.37)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-105.9 to 100.3], Standard Error of Mean 52.06 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -12.9, 95% CI 2-sided [-107.1 to 81.4], Standard Error of Mean 47.52 — Week 52 comparison

34. Secondary Outcome: Mean eGFR at Week 24 and Week 52
Description: The estimated glomerular filtration rate (eGFR) were calculated by the abbreviated Modification of Diet in Renal Disease (MDRD) equation. Adjusted mean difference(treatment-placebo) and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction at Week 24 and Week 52. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments. Only those participants available at the indicated time points were analyzed (represented by n= X, X in the category titles).
Time Frame: Week 24 and Week 52
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: mL/minute/1.73 square meter (m^2)
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 13 | 12
mL/minute/1.73 square meter (m^2)
  Week 24; n=9, 7 | 62.25 (6.119) | 49.33 (6.897)
  Week 52; n= 10, 10 | 58.99 (5.732) | 56.29 (5.765)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -12.92, 95% CI 2-sided [-31.56 to 5.71], Standard Error of Mean 9.440 — Week 24 comparison
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-19.11 to 13.72], Standard Error of Mean 8.315 — Week 52 comparison

35. Secondary Outcome: Mean Prednisolone Use at Week 24
Description: Adjusted mean difference (treatment-placebo) for Prednisolone use and 95% confidence intervals for differences were obtained from MMRM model, with fixed categorical effects of treatment, visit, donor type and treatment-by-visit interaction and fixed continuous covariates of Baseline and Baseline-by-visit interaction at Week 24. A compound symmetry variance structure was used to model the within-participant errors, shared across treatments Only those participants available at indicated timepoints were analyzed (represented by n=X, X in the category titles).
Time Frame: Week 24
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: mg/day
Arm/Group | Placebo | Belimumab 10mg/kg
Number analyzed (Participants) | 10 | 7
mg/day | 5.71 (1.438) | 5.27 (1.713)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-4.84 to 3.96], Standard Error of Mean 2.225

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to 52 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for MITT Population.
Arm/Group | Placebo | Belimumab 10mg/kg
Serious Adverse Events (participants affected / at risk) | 7/13 | 5/12
Other Adverse Events (participants affected / at risk) | 9/13 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Belimumab 10mg/kg (N=12)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal cyst infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Belimumab 10mg/kg (N=12)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (3) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Polyomavirus test positive (Investigations) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epstein-Barr virus test positive (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polyomavirus-associated nephropathy (Infections and infestations) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Ulcerative gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.